CLINICAL TRIAL: NCT01630889
Title: Open-Label Extension Study to Evaluate the Efficacy and Safety of FG-4592 for the Long-Term Maintenance Treatment of Anemia in Dialysis and Non-Dialysis Patients With Chronic Kidney Disease
Brief Title: Open-Label Extension Study for the Long-Term Efficacy and Safety of Roxadustat in Participants With Dialysis and Non-Dialysis Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-059
Record Dates: First submitted 2012-06-08; First posted 2012-06-28 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease; Anemia
Keywords: Kidney; ESRD; End Stage Renal Disease; Anemia; Oral anemia treatment; Hemoglobin levels; Hemodialysis; CKD; Chronic Kidney Disease; Peritoneal; HD; PD; Hb; Erythropoietin; Blood count
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Roxadustat (Experimental): Participants previously randomized to roxadustat will receive roxadustat at the same dose and frequency assigned at the last dose in the previous FibroGen study. Dose adjustments will be implemented (up to a maximum roxadustat dose of 3.0 mg/kg or 400 mg, whichever is lower) every 4 weeks to maintain Hb levels at 10.0-12 grams (g)/deciliter (dL). However, if a participant, at any dose, experiences an event of excessive hematopoiesis then the participant's dose will be immediately reduced, or an event of rapidly declining Hb then the participant's dose will be immediately increased. Participants will be permitted to receive roxadustat for up to 8 years.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Oral capsule
  Other Names: FG-4592

SUMMARY:
The purpose of this open-label extension study is to evaluate long-term efficacy and safety of roxadustat in maintaining hemoglobin (Hb) in participants with dialysis and non-dialysis chronic kidney disease (CKD) who have completed the Treatment Period of a roxadustat FibroGen-sponsored anemia study.

DETAILED DESCRIPTION:
This is an open-label, long-term maintenance study of roxadustat anemia therapy in participants with dialysis and non-dialysis CKD who have completed the Treatment Period of a roxadustat FibroGen-sponsored anemia study. Participants assigned to roxadustat in the previous study will continue to receive the same roxadustat dose and dosing frequency, unless a dose adjustment is required.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age 18 years
2. Completed the Treatment Period of an ongoing roxadustat FibroGen-sponsored anemia study in the United States.

Exclusion Criteria

1. Participants assigned to epoetin alfa in a previous ongoing roxadustat anemia study
2. Pregnant or breastfeeding females
3. Females of childbearing potential, unless using adequate contraception; male participants with sexual partners of childbearing potential who are not on birth control unless the male participant agrees to use adequate contraception
4. Participants who received roxadustat in a previous study that did not demonstrate adequate hemoglobin response per the investigator's clinical judgment
5. Any medical condition that in the opinion of the investigator may pose a safety risk to a participant in this study or which may interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peony Yu, Study Director — Kyntra Bio
Locations (7):
- United States (4):
  - APEX Research, Riverside, California
  - Greenbelt, Maryland
  - Mountain Kidney & HTN Associates, PA, Asheville, North Carolina
  - Arlington Nephrology, Arlington, Texas
- Puerto Rico (3):
  - Consolidated Medical Plaza, Caguas
  - CAIMED School of Medicine, Ponce
  - San Juan

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Roxadustat: Participants previously randomized to roxadustat received roxadustat at the same dose and frequency assigned at the last dose in the previous FibroGen study. Dose adjustments were implemented (up to a maximum roxadustat dose of 3.0 mg/kg or 400 mg, whichever is lower) every 4 weeks to maintain Hb levels at 10.0-12 grams (g)/deciliter (dL). However, if a participant, at any dose, experienced an event of excessive hematopoiesis then the participant's dose was immediately reduced, or an event of rapidly declining hemoglobin (Hb) then the participant's dose was immediately increased. Participants were permitted to receive roxadustat for up to 8 years.
Period: Overall Study
Arm/Group | Roxadustat
Started | 15
Received at Least 1 Dose of Study Drug | 15
Completed | 5
Not Completed | 10
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other than Specified | 2
Not completed — Lost to Follow-up | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Groups:
- Roxadustat: Participants previously randomized to roxadustat received roxadustat at the same dose and frequency assigned at the last dose in the previous FibroGen study. Dose adjustments were implemented (up to a maximum roxadustat dose of 3.0 mg/kg or 400 mg, whichever is lower) every 4 weeks to maintain Hb levels at 10.0-12 g/dL. However, if a participant, at any dose, experienced an event of excessive hematopoiesis then the participant's dose was immediately reduced, or an event of rapidly declining Hb then the participant's dose was immediately increased. Participants were permitted to receive roxadustat for up to 8 years.
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hb Over Time
Description: Hb baseline was defined as the mean of the central laboratory Hb value from the baseline visit at Day 1 (prior to receiving the first dose of study drug in this study), plus any other central lab Hb values within 15 days prior to Day 1 regardless of fasting. The specific duration over which the participants were assessed was identified as "over time" for the endpoint in the study protocol. Therefore, to be consistent with the endpoint in the study protocol, an individual timepoint was not identified for this primary outcome measure.
Time Frame: Baseline, Weeks 8, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 252, 264, 288, 312, 336, 360, and 384
Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
g/dL
  Baseline | 10.05 (0.931)
  Change at Week 8: number analyzed (Participants) | 14
  Change at Week 8 | 1.26 (0.633)
  Change at Week 24: number analyzed (Participants) | 13
  Change at Week 24 | 1.58 (0.959)
  Change at Week 48: number analyzed (Participants) | 14
  Change at Week 48 | 1.94 (1.324)
  Change at Week 72: number analyzed (Participants) | 11
  Change at Week 72 | 2.54 (1.234)
  Change at Week 96: number analyzed (Participants) | 8
  Change at Week 96 | 1.18 (1.141)
  Change at Week 120: number analyzed (Participants) | 8
  Change at Week 120 | 1.61 (0.815)
  Change at Week 144: number analyzed (Participants) | 7
  Change at Week 144 | 1.96 (0.804)
  Change at Week 168: number analyzed (Participants) | 6
  Change at Week 168 | 1.40 (1.441)
  Change at Week 192: number analyzed (Participants) | 6
  Change at Week 192 | 1.02 (1.063)
  Change at Week 216: number analyzed (Participants) | 5
  Change at Week 216 | 1.34 (1.062)
  Change at Week 240: number analyzed (Participants) | 5
  Change at Week 240 | 1.02 (0.779)
  Change at Week 264: number analyzed (Participants) | 4
  Change at Week 264 | 1.63 (1.640)
  Change at Week 288: number analyzed (Participants) | 4
  Change at Week 288 | 0.00 (1.647)
  Change at Week 312: number analyzed (Participants) | 3
  Change at Week 312 | 0.23 (0.416)
  Change at Week 336: number analyzed (Participants) | 2
  Change at Week 336 | 0.70 (0.000)
  Change at Week 360: number analyzed (Participants) | 1
  Change at Week 360 | -1.20 (NA) — NA=Standard Deviation cannot be calculated with N of 1.
  Change at Week 384: number analyzed (Participants) | 1
  Change at Week 384 | -0.40 (NA) — NA=Standard Deviation cannot be calculated with N of 1.

2. Secondary Outcome: Number of Participants With Hb ≥10 g/dL
Description: Hb baseline was defined as the mean of the central laboratory Hb value from the baseline visit at Day 1 (prior to receiving the first dose of study drug in this study), plus any other central lab Hb values within 15 days prior to Day 1 regardless of fasting.
Time Frame: Baseline up to Week 384
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
Participants
  Baseline | 9
  Week 8 | 13
  Week 24 | 13
  Week 48 | 13
  Week 72 | 11
  Week 96 | 7
  Week 120 | 8
  Week 144 | 7
  Week 168 | 5
  Week 192 | 5
  Week 216 | 5
  Week 240 | 5
  Week 264 | 4
  Week 288 | 3
  Week 312 | 3
  Week 336 | 2
  Week 360 | 1
  Week 384 | 1

3. Secondary Outcome: Number of Participants Receiving Rescue Therapy (Composite of Blood Transfusions, Intravenous [IV] Iron, Erythropoiesis-Stimulating Agent [ESA])
Time Frame: Baseline up to Week 385
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
Participants
  Blood Transfusion | 1
  IV Iron | 5
  ESA | 1
  No Rescue Therapy | 8

4. Secondary Outcome: Mean Weekly Dose of Study Drug Over Time
Description: Weekly dose amount was the actual total dose amounts within a week, windowed by 7-day period from Day 1. The mean weekly dose is presented for selected time periods based on timepoints reported in Outcome Measures 1 and 2.
Time Frame: Baseline up to Week 384
Population: Participants who received at least 1 dose of study drug. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
mg
  Week 1-4 | 257.0 (140.33)
  Week 5 - 8: number analyzed (Participants) | 14
  Week 5 - 8 | 252.4 (115.26)
  Week 21 - 24: number analyzed (Participants) | 13
  Week 21 - 24 | 282.3 (218.07)
  Week 41 - 48: number analyzed (Participants) | 14
  Week 41 - 48 | 318.4 (216.90)
  Week 61 - 72: number analyzed (Participants) | 11
  Week 61 - 72 | 236.7 (108.57)
  Week 85 - 96: number analyzed (Participants) | 8
  Week 85 - 96 | 155.9 (114.27)
  Week 109 - 120: number analyzed (Participants) | 8
  Week 109 - 120 | 142.8 (105.10)
  Week 133 - 144: number analyzed (Participants) | 8
  Week 133 - 144 | 140.3 (101.03)
  Week 157 - 168: number analyzed (Participants) | 6
  Week 157 - 168 | 152.2 (111.19)
  Week 181 - 192: number analyzed (Participants) | 6
  Week 181 - 192 | 195.6 (184.77)
  Week 205 - 216: number analyzed (Participants) | 6
  Week 205 - 216 | 209.4 (156.13)
  Week 229 - 240: number analyzed (Participants) | 5
  Week 229 - 240 | 225.7 (164.58)
  Week 253 - 264: number analyzed (Participants) | 4
  Week 253 - 264 | 327.9 (169.82)
  Week 277 - 288: number analyzed (Participants) | 4
  Week 277 - 288 | 324.0 (190.75)
  Week 301 - 312: number analyzed (Participants) | 4
  Week 301 - 312 | 319.2 (196.98)
  Week 325 - 336: number analyzed (Participants) | 3
  Week 325 - 336 | 413.3 (180.37)
  Week 349 - 360: number analyzed (Participants) | 2
  Week 349 - 360 | 389.6 (156.15)
  Week 373 - 384: number analyzed (Participants) | 1
  Week 373 - 384 | 250.0 (NA) — NA=Standard Deviation cannot be calculated with N of 1.

5. Secondary Outcome: Number of Participants With Dose Adjustments up to Week 52
Description: Dose adjustments include dose increases, dose interruptions, and dose reductions.
Time Frame: Baseline up to Week 52
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
Participants
  Participants without Change | 1
  Participants with 1 Dose Increase | 5
  Participants with 2 Dose Increases | 1
  Participants with >2 Dose Increases | 6
  Participants with 1 Dose Interruption | 1
  Participants with 2 Dose Interruptions | 1
  Participants with >2 Dose Interruptions | 0
  Participants with 1 Dose Reduction | 2
  Participants with 2 Dose Reductions | 8
  Participants with >2 Dose Reductions | 2

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical event in a participant who received study drug whether or not the event is considered drug related. TEAEs were defined as any event that either began or worsened after the first administration of study drug and within 28 days of the last dose. Serious AE criteria included death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed here. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 385
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 15
Participants
  Any TEAEs | 14
  Serious TEAEs | 9

ADVERSE EVENTS:
Time Frame: Baseline up to Week 385
Description: Participants who received at least 1 dose of study drug.
Arm/Group | Roxadustat
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=15)
Hemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Ventricular fibrillation (Cardiac disorders) | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Renal tubular necrosis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Shock hemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Roxadustat (N=15)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Cataract (Eye disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Injection site rash (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Abdominal infection (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Chikungunya virus infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 1/10 — This is a sex-specific adverse event that only affects female participants.
Viral upper respiratory tract infection (Infections and infestations) | 3
Vulvovaginal candidiasis (Infections and infestations) | 1/10 — This is a sex-specific adverse event that only affects female participants.
Bone contusion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2
Blood pressure increased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Thrombosis in device (Product Issues) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1/10 — This is a sex-specific adverse event that only affects female participants.
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/10 — This is a sex-specific adverse event that only affects female participants.
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Loss of personal independence in daily activities (Social circumstances) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen.

The investigator can only publish after the multisite consortium publishes (or tries to publish and fails).

FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT01630889/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT01630889/SAP_001.pdf